CLINICAL TRIAL: NCT04698577
Title: Evaluation of a School-Based Attention Training Programme for Improving Sustained Attention: A Cluster Randomised Pilot Study
Brief Title: Evaluation of a School-Based Attention Training Programme for Improving Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Principal Investigator, Eadaoin Slattery, Ms., University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_10_10_EHS
Record Dates: First submitted 2020-12-23; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Attention Concentration Difficulty
Keywords: Attention training; Cognitive training; Attention; Sustained attention; Working memory; School intervention; Children

STUDY DESIGN:
Intervention Model Description: This is a two arm, single-blind, pilot cluster randomised study. Participants were randomly allocated to the attention training group or active control group based on class groups (three class groups of fourth-class students and one class group of fifth-class students).
Who Masked: Participant
Masking Description: Participants and their parents were blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Training (Experimental): Engaged in sustained updating by mentally keeping score during an interactive game without written or verbal aids.
  Participants received 15-minute sessions, three times a week for six weeks (18 sessions in total).
  Interventions: Behavioral: Attention Training
- Active Control (Active Comparator): Played the same interactive game as the attention training group without the requirement of mentally keeping score.
  Participants received 15-minute sessions, three times a week for six weeks (18 sessions in total).
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Attention Training — The training was delivered face-to-face in groups of three participants. Participants were involved in a game of table tennis with two players and one spectator. The roles were rotated every 5 minutes so that each participant experienced 10 minutes of play and 5 minutes of observation. The game was played as normal with one point awarded to the player for every score achieved. All 3 players were asked to keep the score of the game in their minds during each 5-minute round. Participants had two objectives 1) to play and win the game and 2) to silently keep the score of the game. The researcher watched the game and accurately kept score, using a notepad. At the end of every 5-minute round, the researcher paused play and asked each child to write down the score they were holding in their mind. The researcher then revealed the true score, asked participants to swap roles and commence another round.
  Arms: Attention Training
Behavioral: Active Control — The control group was the same as the training group except for the core training mechanism; children were not required to mentally keep score. The researcher kept score by continually calling out the updated score as each point was won. The observing child was simply told to wait his/her turn.
  Arms: Active Control

SUMMARY:
This study evaluates a school-based attention training programme for improving sustained attention in children.

DETAILED DESCRIPTION:
Sustained attention is an elementary attentional function that is essential for effective learning and functioning in school. Poor sustained attention is a relatively common problem in childhood with as many as 24% of children exhibiting frequent inattention. Children with attentional difficulties are at increased risk for a variety of negative educational outcomes, including lower standardised grades, dropping out of school and repeating a year. This evidence highlights the need to develop interventions aimed at enhancing students' sustained attention capacity. Current school-based interventions for student attention problems include intervention strategies targeting behavioural, academic and self-regulation. However, none of these interventions aim to enhance attentional capacity. Attention network training (or attention training) has been identified as a potentially promising intervention for enhancing attentional capacity. This pilot study aimed to evaluate the preliminary efficacy of a theory-driven attention training programme, Keeping Score!, in improving students' capacity to sustain attention in a school setting. Training was based on sustained updating. Children engaged this process by mentally keeping score during an interactive face-to-face game without external aids. The study used a cluster randomised design. Students (N = 36) were assigned based on their class group to either the 6-week attention training programme (n = 18) or an active control (n = 18). Outcome measures were assessed at baseline, immediately after training and an approximate 6-week follow up.

ELIGIBILITY:
Inclusion Criteria:

* 4th and 5th class students
* aged 9 to 11 years
* parent consent and participant assent

Exclusion Criteria:

-

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Vigil subtest of the Test of Everyday Attention for Children - Second Edition (TEA-Ch2). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Vigil subtest of the TEA-Ch2 is a measure of sustained attention. Participants were required to count slow, irregularly paced stimuli. Participants completed 10 trials. The outcome variable was the total number of correct trials. Higher scores indicate a better outcome.
Change in scores on the Cerberus subtest of the Test of Everyday Attention for Children - Second Edition (TEA-Ch2). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Cerberus subtest of the TEA-Ch2 is a measure of sustained attention. Participants were required to listen to short clips and respond (press the spacebar) to a target auditory stimulus while ignoring other sounds. Participants completed 15 trials. The outcome measure was mean reaction time in msecs weighted for accuracy. Lower scores indicate a better outcome.
Change in scores on the Sustained Attention to Response Task (SART) subtest of the Test of Everyday Attention for Children - Second Edition (TEA-Ch2). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The SART subtest of the TEA-Ch2 is a measure of sustained attention. Participants were required to respond (press the spacebar) to every shape (go-trial) that appeared on screen but not to respond to a triangle (no-go trial). There were 20 no-go trials. The outcome measure was errors of commission (no-go trial responses). Lower scores indicate a better outcome.

SECONDARY OUTCOMES:
Change in scores on the Digit Span Backwards subtest of the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Digit Span Backwards subtest is a measure of working memory. Participants were required to repeat a dictated string of numbers in the reverse order. The task was discontinued when the participant failed to answer both trials of a set correctly. The outcome measure was the total number of correctly recalled trials. The maximum total score is 18. Higher scores indicate a better outcome.
Change in scores on the Operation Span subtest of the Adaptive Composite Complex Span (ACCES). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Operation Span subtest is a measure of working memory. Participants were required to evaluate maths problems while memorising letters. Participants completed 6 trials. The number of stimulus-problem pairs within a trial varied between two and eight. The outcome measure was the total number of stimuli correctly recalled. Higher scores indicate a better outcome.
Change in scores using the Symmetry Span subtest of the Adaptive Composite Complex Span (ACCES). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Symmetry Span subtest is a measure of working memory. Participants were required to evaluate whether geometric shapes were symmetrical while remembering spatial locations. Participants completed 6 trials. The number of stimulus-problem pairs within a trial varied between two and eight. The outcome measure was the total number of stimuli correctly recalled. Higher scores indicate a better outcome .
Change in scores on the Digit Span Forward subtest of the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The Digit Span Forwards subtest is a measure of short-term memory. Participants were required to repeat a dictated string of numbers in the same order. The task was discontinued when the participant failed to answer both trials of a set correctly. The outcome measure was the total number of correctly recalled trials. The maximum total score is 18. Higher scores indicate a better outcome.
Change in parent ratings of executive function behaviour on the Behaviour Rating Inventory of Executive Function - Second Edition (BRIEF-2). | Baseline (pre-training), post-training at approximately 6 weeks after baseline and study completion at approximately 12 weeks after baseline.
  The BRIEF-2 assesses everyday behaviours associated with executive function in the home environment. Parents rated 63 items on a three-point Likert scale (0 = never, 1 = sometimes and 2 = often). The following indices were used: Behaviour Regulation Index (BRI), Emotion Regulation Index (ERI), Cognitive Regulation Index (CRI) and Global Executive Composite (GEC). Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eadaoin J Slattery, M.Sc., Principal Investigator — University of Limerick; Laura P McAvinue, PhD, Study Director — University College Dublin / University of Limerick; Patrick Ryan, D.Clin.Psych, Study Director — University of Limerick; Donal G Fortune, PhD, Study Director — University of Limerick
Locations (1):
- Department of Psychology, University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The anonymised dataset is available on the Open Science Framework (OSF).
Supporting Information: Analytic Code
Time Frame: Available from 23/11/2020
Access Criteria: Data is publicly available
URL: https://osf.io/7axwr/

REFERENCES:
- [Background] Gonthier C, Aubry A, Bourdin B. Measuring working memory capacity in children using adaptive tasks: Example validation of an adaptive complex span. Behav Res Methods. 2018 Jun;50(3):910-921. doi: 10.3758/s13428-017-0916-4. PMID 28643158
- [Background] Dopfner M, Breuer D, Wille N, Erhart M, Ravens-Sieberer U; BELLA study group. How often do children meet ICD-10/DSM-IV criteria of attention deficit-/hyperactivity disorder and hyperkinetic disorder? Parent-based prevalence rates in a national sample--results of the BELLA study. Eur Child Adolesc Psychiatry. 2008 Dec;17 Suppl 1:59-70. doi: 10.1007/s00787-008-1007-y. PMID 19132305
- [Background] DuPaul GJ, Gormley MJ, Laracy SD. School-based interventions for elementary school students with ADHD. Child Adolesc Psychiatr Clin N Am. 2014 Oct;23(4):687-97. doi: 10.1016/j.chc.2014.05.003. Epub 2014 Aug 1. PMID 25220080
- [Background] Tang YY, Posner MI. Attention training and attention state training. Trends Cogn Sci. 2009 May;13(5):222-7. doi: 10.1016/j.tics.2009.01.009. Epub 2009 Apr 16. PMID 19375975